CLINICAL TRIAL: NCT03031535
Title: A Two-Part, Phase 1, Randomized, Crossover Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intranasal Octreotide (DP1038) Versus Subcutaneous Sandostatin® Injection in Healthy Adult Volunteers
Brief Title: Study of Intranasal Octreotide (DP1038) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dauntless Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP1038-PK-101
Record Dates: First submitted 2017-01-17; First posted 2017-01-25 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-01

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Intervention Model Description: This study consists of two study parts. In Study Part 1, 12 subject will be randomized into one of four study arms using a 4x4 modified latin square design.
  In Study Part 2, subjects will be randomized into one of two arms using a 2x2 crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Study Part 1 - Arm 1 (Experimental): Day 1 - Intranasal octreotide acetate (DP1038) - 400 micrograms; Day 3 - Intranasal octreotide acetate (DP1038) - 1200 micrograms; Day 5 - Intranasal octreotide acetate (DP1038) - 2000 micrograms; Day 7 - Subcutaneous octreotide acetate (Sandostatin Injection) - 100 micrograms.
  Interventions: Drug: Intranasal octreotide acetate; Drug: Subcutaneous octreotide acetate
- Study Part 1 - Arm 2 (Experimental): Day 1 - Intranasal octreotide acetate (DP1038) - 1200 micrograms; Day 3 - Intranasal octreotide acetate (DP1038) - 400 micrograms; Day 5 - Subcutaneous octreotide acetate (Sandostatin Injection) - 100 micrograms; Day 7 - Intranasal octreotide acetate (DP1038) - 2000 micrograms.
  Interventions: Drug: Intranasal octreotide acetate; Drug: Subcutaneous octreotide acetate
- Study Part 1 - Arm 3 (Experimental): Day 1 - Intranasal octreotide acetate (DP1038) - 2000 micrograms; Day 3 - Subcutaneous octreotide acetate (Sandostatin Injection) - 100 micrograms; Day 5 - Intranasal octreotide acetate (DP1038) - 400 micrograms; Day 7 - Intranasal octreotide acetate (DP1038) - 1200 micrograms.
  Interventions: Drug: Intranasal octreotide acetate; Drug: Subcutaneous octreotide acetate
- Study Part 1 - Arm 4 (Experimental): Day 1 - Subcutaneous octreotide acetate (Sandostatin Injection) - 100 micrograms; Day 3 - Intranasal octreotide acetate (DP1038) - 2000 micrograms; Day 5 - Intranasal octreotide acetate (DP1038) - 1200 micrograms; Day 7 - Intranasal octreotide acetate (DP1038) - 400 micrograms.
  Interventions: Drug: Intranasal octreotide acetate; Drug: Subcutaneous octreotide acetate
- Study Part 2 - Arm 1 (Experimental): Day 1 - 1 microgram/kilogram of growth hormone-releasing hormone (GHRH) + 30 grams arginine hydrochloride; Day 3 - Intranasal octreotide acetate (DP1038) - dose to be determined from Study Part 1 PK results + 1 microgram/kilogram of GHRH + 30 grams arginine hydrochloride; Day 5 - SC octreotide acetate (Sandostatin Injection) 100 micrograms + 1 microgram/kilogram of GHRH + 30 grams arginine hydrochloride.
  Interventions: Drug: Intranasal octreotide acetate; Drug: Subcutaneous octreotide acetate; Diagnostic Test: Growth hormone-releasing hormone; Diagnostic Test: Arginine hydrochloride
- Study Part 2 - Arm 2 (Experimental): Day 1 - 1 microgram/kilogram of GHRH + 30 grams arginine hydrochloride; Day 3 - SC octreotide acetate (Sandostatin Injection) 100 micrograms + 1 microgram/kilogram of GHRH + 30 grams arginine hydrochloride; Day 5 - Intranasal octreotide acetate (DP1038) - dose to be determined from Study Part 1 PK results + 1 microgram/kilogram of GHRH + 30 grams arginine hydrochloride.
  Interventions: Drug: Intranasal octreotide acetate; Drug: Subcutaneous octreotide acetate; Diagnostic Test: Growth hormone-releasing hormone; Diagnostic Test: Arginine hydrochloride

INTERVENTIONS:
Drug: Intranasal octreotide acetate — Intranasal spray of octreotide acetate
  Other Names: DP1038
Drug: Subcutaneous octreotide acetate — Subcutaneous injectable solution of octreotide acetate
  Other Names: Sandostatin Injection
Diagnostic Test: Growth hormone-releasing hormone — Part of the well established GHRH/Arginine challenge to detect GH deficiency.
  Other Names: GHRH
  Arms: Study Part 2 - Arm 1; Study Part 2 - Arm 2
Diagnostic Test: Arginine hydrochloride — Part of the well established GHRH/Arginine challenge to detect GH deficiency.
  Other Names: R-Gene 10
  Arms: Study Part 2 - Arm 1; Study Part 2 - Arm 2

SUMMARY:
The purpose of the study is to investigate the drug octreotide acetate in a new intranasal formulation and compare it to the FDA-approved subcutaneous (SC) injection formulation. The two octreotide acetate formulations will be evaluated following separate administrations for safety and tolerability including any side effects, the speed at which the drug is absorbed and eliminated in the body, and the ability of the drug to lower the levels of growth hormone (GH) and insulin-like growth factor 1 (IGF-1).

DETAILED DESCRIPTION:
Octreotide is a synthetic octapeptide analog of naturally occurring somatostatin, with similar pharmacological effects but a longer duration of action. It inhibits the pathological secretion of GH from pituitary adenomas, and of serotonin and other hormones by tumors of the gastroenteropancreatic endocrine system. Currently, only injectable octreotide and somatostatin analogs have been approved, for the indications of acromegaly, carcinoid tumors, and vasoactive intestinal peptide tumors.

DP1038, an intranasal formulation of octreotide, is being developed for the treatment of acromegaly, a rare chronic disorder arising from the overproduction of GH, predominantly by pituitary adenomas. Excess GH and associated IGF-1 levels are responsible for multiple symptoms (e.g., headache, tissue swelling, perspiration, joint pain) and significant comorbidities (e.g., diabetes, sleep apnea, cardiovascular abnormalities such as hypertension). In most patients with acromegaly, octreotide consistently normalizes GH and IGF-1 serum concentrations, thereby markedly reducing clinical symptoms.

ELIGIBILITY:
Key eligibility criteria:

Inclusion Criteria:

* Body mass index (BMI) 18 and <28 kg/m2 (to minimize variability in SC absorption).
* Be in good general health.

Exclusion Criteria:

* Use of any tobacco product within 30 days prior to first dose of study drug.
* Use of any prescription or non-prescription drugs or dietary supplements within 7 days, insulin or hypoglycemic drugs within 3 months, estrogen-containing medication within 3 months, or drugs that may affect GH and IGF-1 levels (e.g., alpha-adrenergic, beta-adrenergic, and cholinergic drugs) within 1 month prior to dosing.
* Subjects will also be excluded if they have a history of gallbladder disease, hypothyroidism, or unexplained hypoglycemia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects reporting adverse events (AEs)/serious adverse events (SAEs). | Both Study Parts: Entire study duration, an average of 1 week.
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  AUC from pre-dose to time 't' (AUC[0-t]) and pre-dose to infinite time (AUC[0-infinity]) of intranasal DP1038 versus subcutaneous Sandostatin Injection.
Maximum plasma concentration (Cmax) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  Maximum octreotide plasma concentration (Cmax) of intranasal DP1038 versus subcutaneous Sandostatin Injection.
Time to maximum plasma concentration (Tmax) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  Time to maximum octreotide plasma concentration (Tmax) of intranasal DP1038 versus subcutaneous Sandostatin Injection.
Lagtime (Tlag) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  Tlag is the amount of time required to obtain the first measurable concentration of plasma octreotide.
Terminal elimination half-life (t1/2) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  Plasma decay half-life is the time measured for the octreotide plasma concentration to decrease by one half.
Apparent systemic clearance (CL/F) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  CL/F is the volume of plasma cleared of octreotide per unit time.
Elimination rate constant (lambda z) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  Lambda z is a quantitative measure of the rate at which octreotide is removed from the body.
Apparent volume of distribution (Vz/F) | Part 1 - Days 1, 3, 5, and 7 & Part 2 - Days 3 and 5: Pre-dose, 5 min, 10 min, 20 min, 30 min, 40 min, 1 hr, 2 hr, 4 hr, and 8 hr post-dose.
  Vz/F is the apparent volume of distribution of octreotide during the terminal elimination phase not corrected for bioavailability.
Growth hormone (GH) concentrations over time. | Part 2 only - Days 1, 3, and 5: -60 min, -40 min, -20 min, and -5 min pre-dose and post-arginine infusion completion at 0 min, 20 min, 40 min, 60 min, 80 min, 100 min, 120 min, 140 min, and 160 min, and at 4 and 8 hr.
  GH levels will be collected over time to compare the suppressive ability of intranasal octreotide (DP1038) versus subcutaneous octreotide (Sandostatin Injection) compared to no octreotide on the GH levels after a GHRH/arginine challenge.
Insulin-like growth factor-1 (IGF-1) concentrations over time. | Part 2 only - Days 1, 3, and 5: -60 min, -40 min, -20 min, and -5 min pre-dose and post-arginine infusion completion at 0 min, 20 min, 40 min, 60 min, 80 min, 100 min, 120 min, 140 min, and 160 min, and at 4 and 8 hr.
  IGF-1 levels will be collected over time to compare the suppressive ability of intranasal octreotide (DP1038) versus subcutaneous octreotide (Sandostatin Injection) compared to no octreotide on IGF-1 levels after a GHRH/arginine challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zacher, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No